CLINICAL TRIAL: NCT02606071
Title: Italian Registry On Multipoint Left Ventricular
Brief Title: Italian Registry On Multipoint Left Ventricular Pacing
Acronym: IRON-MPP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Giovanni B Forleo, MD, Luigi Sacco University Hospital
Other Study IDs: MPP04
Record Dates: First submitted 2015-11-06; First posted 2015-11-17 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Heart Failure; Ventricular Fibrillation; Ventricular Tachycardia
Keywords: cardiac resynchronization therapy; multipoint left ventricular pacing
MeSH Terms: conditions — Heart Failure; Ventricular Fibrillation; Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: CRT-D — HF patients treated in clinical practice with a CRT-D device

SUMMARY:
The IRON-MPP is a prospective multicenter, observational registry designed to collect clinical and device data from a large cohort of HF patients treated in clinical practice with a CRT-D device with the ability to deliver Multi Point Pacing.

The purpose of the Registry is to collect data on how MPP-devices are being used by physicians in order to better understand how to improve the clinical care of patients and effectiveness of MPP therapy.

ELIGIBILITY:
Inclusion Criteria:

- Patients implanted with a St. Jude Medical CRT-D system with MPP capability

Exclusion Criteria:

- Patients currently participating in any other clinical investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HF patients treated in clinical practice with a CRT-D device with the ability to deliver MPP
Sampling Method: Non-Probability Sample
Enrollment: 436 (Actual)
Dates: Start 2013-08; Primary Completion 2016-09 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | 6 Months
  Changes in Left ventricular ejection fraction

SECONDARY OUTCOMES:
Heart Failure Hospitalizations | 12 months
Appropriate device interventions | 12 months
  Number of participants with appropriate device interventions (anti-tachycardia pacing or shock)
Echocardiographic changes | 12 months
  Left ventricular end systolic volume
QRS Duration | Baseline and six months
  Changes in QSR duration between MPP and conventional biventricular pacing

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Forleo, Principal Investigator — Policlinico Tor Vergata
Locations (3):
- Italy (3):
  - Ospedale Santa Maria della Misericordia, Rovigo
  - Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Ospedale Maria Vittoria, Torino

REFERENCES:
- [Derived] Forleo GB, Santini L, Giammaria M, Potenza D, Curnis A, Calabrese V, Ricciardi D, D'agostino C, Notarstefano P, Ribatti V, Morani G, Mantica M, Di Biase L, Bertaglia E, Calo L, Zanon F. Multipoint pacing via a quadripolar left-ventricular lead: preliminary results from the Italian registry on multipoint left-ventricular pacing in cardiac resynchronization therapy (IRON-MPP). Europace. 2017 Jul 1;19(7):1170-1177. doi: 10.1093/europace/euw094. PMID 27189954